CLINICAL TRIAL: NCT00575146
Title: Ketogenic Diet for Patients With Recurrent Glioblastoma
Brief Title: Ketogenic Diet for Recurrent Glioblastoma
Acronym: ERGO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Evomed MedizinService GmbH (Unknown)
Responsible Party: Principal Investigator, J. Rieger, Dr. Johannes Rieger, University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERGO
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Recurrent Glioblastoma
Keywords: glioblastoma; ketogenic diet
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): ketogenic diet
  Interventions: Dietary Supplement: TAVARLIN

INTERVENTIONS:
Dietary Supplement: TAVARLIN — ketogenic diet, dietary supplementary products provided by TAVARLIN

SUMMARY:
To determine whether a mild ketogenic diet can influences quality of life and survival of patients with recurrent glioblastoma

DETAILED DESCRIPTION:
Increased glycolysis and reduced oxidative phosphorylation is a characteristic property of many tumors. A change of nutrition by limiting carbohydrates and increasing the proportion of fatty acids and proteins can lead to ketogenic metabolism and might limit energy production in tumor cells and therefore inhibit tumor growth. Standard treatment for glioblastoma includes resection, irradiation and temozolomide chemotherapy. If there is tumor recurrence, no standard therapy is established. Therapeutic options in this situation include resection, irradiation or another chemotherapy. However, some patients cannot be treated in this situation, because none of the available treatment options seems reasonable or applicable, for example if no additional chemotherapy can be started at the time of recurrence due to myelosuppression. The pilot study examines whether in this situation a ketogenic diet can be applied to the patients and may inhibit tumor growth and influence the quality of life of the patients.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* histological diagnosis of glioblastoma or gliosarcoma
* on MRI measurable tumor
* interval of at least 6 months after primary resection
* completed radiotherapy, interval of at least 3 months after completion of radiotherapy
* relapse during or after temozolomide chemotherapy, other chemotherapy not possible, not reasonable or not wanted by the patient
* Karnofsky-Index >= 60%, ECOG <= 2
* life expectancy of at least 12 weeks
* creatinine <= 1.5 mg/dl, urea <= 50 mg/dl
* INR <= 1,5, GOT <= 7 x of normal value, GPT <= 7 x of normal value

Exclusion Criteria:

* bowel obstruction or subileus
* diabetes mellitus, HbA1c > 6,1 %
* heart failure (NYHA > 2), myocardial infarction within the last 6 months, atrial fibrillation
* acute infection
* conditions that may strongly reduce compliance to the diet or increase risk of the diet
* dementia or clinically relevant alterations of the mental state which interfere with the applicability of the diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Rieger, MD, Principal Investigator — Senckenberg Institute of Neurooncology, University of Frankfurt
Locations (2):
- Germany (2):
  - Senckenberg Institute of Neurooncology, Frankfurt
  - Department of General Neurology and Hertie-Institute of Clinical Brain Research, University of Tuebingen, Tübingen

REFERENCES:
- [Result] Rieger J, Bahr O, Maurer GD, Hattingen E, Franz K, Brucker D, Walenta S, Kammerer U, Coy JF, Weller M, Steinbach JP. ERGO: a pilot study of ketogenic diet in recurrent glioblastoma. Int J Oncol. 2014 Jun;44(6):1843-52. doi: 10.3892/ijo.2014.2382. Epub 2014 Apr 11. PMID 24728273

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketogenic Diet: unrestricted ketogenic diet (< 50-60 g carbohydrates per day) and dietary supplementary products provided by Tavarlin
Period: Overall Study
Arm/Group | Ketogenic Diet
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Ketogenic Diet: ketogenic diet
Arm/Group | Ketogenic Diet
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Number; unit: participants]
  Germany | 20

OUTCOME MEASURES:

1. Primary Outcome: Applicability as Measured by Discontinuation of Study Treatment Due to Intolerability
Description: percentage of patients who discontinued diet due to intolerability
Time Frame: until progression for up to 12 months
Measure: Number; unit: percent of participants
Groups:
- Ketogenic Diet: unrestricted ketogenic diet
Arm/Group | Ketogenic Diet
Number analyzed (Participants) | 20
percent of participants | 15

2. Secondary Outcome: Progression-free-survival
Description: measured by Macdonald-Criteria
Time Frame: until progression for up to 12 months
Population: for the analyis of PFS and OS, 3 patients who discontinued the diet in the absence of progression were excluded
Measure: Median (Full Range); unit: weeks
Arm/Group | Ketogenic Diet
Number analyzed (Participants) | 17
weeks | 5 [3 to 13]

3. Secondary Outcome: Overall Survival
Description: Participants were followed until reported death or last contact until 05/2011
Time Frame: death/last contact, an average of about 1 year
Measure: Median (Full Range); unit: weeks
Arm/Group | Ketogenic Diet
Number analyzed (Participants) | 20
weeks | 32 [6 to 159]

4. Secondary Outcome: Frequency of Seizures
Time Frame: while on study treatment for up to 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Ketosis
Time Frame: while on study treatment for up to 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Quality of Life
Time Frame: while on study treatment for up to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ketogenic Diet
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Because of the small number of patients efficacy cannot be concluded by the results of the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No